CLINICAL TRIAL: NCT01114165
Title: Value of the LightCycler® SeptiFast Test MGRADE for the Pathogen Detection in Neutropenic Hematological Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Pfizer (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UKM-SF-042010
Record Dates: First submitted 2010-04-23; First posted 2010-05-03 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-11

CONDITIONS: Hematologic Diseases; Neutropenia; Febrile Neutropenia; Sepsis
Keywords: Neutropenia; Febrile Neutropenia; Sepsis; Polymerase Chain Reaction
MeSH Terms: conditions — Hematologic Diseases; Neutropenia; Febrile Neutropenia; Sepsis

ARMS (2):
- SeptiFast Test (Experimental): Pathogen detection by SeptiFast Test as an adjunct to traditional microbiological assessments including blood culture
  Interventions: Other: Detection of microbial DNA in blood by SeptiFast Test
- Only Conventional Diagnostics (Active Comparator): Pathogen detection only by conventional microbiological assessments, e.g. blood culture
  Interventions: Other: Pathogen detection by blood culture

INTERVENTIONS:
Other: Detection of microbial DNA in blood by SeptiFast Test — The SeptiFast Test is a multiplex polymerase chain reaction (PCR) test that can detect nucleic acids from the most common pathogens (approximately 90%) responsible for hospital-associated bacteremia and takes approx. 6 hours to perform
  Arms: SeptiFast Test
Other: Pathogen detection by blood culture — Blood culture is a conventional microbiological method of pathogen detection. Results from blood cultures are usually not available until 24 to 72 hours after sampling
  Arms: Only Conventional Diagnostics

SUMMARY:
The overall objective of this study is to assess the clinical value of the SeptiFast Test as an adjunct to traditional microbiological, clinical, and other laboratory assessments in early detection and identification of a potential pathogen and therefore early targeted antimicrobial management of neutropenic hematological patients with suspected infection or sepsis.

DETAILED DESCRIPTION:
Infections, including sepsis, continue to be a major cause of morbidity and mortality in patients with hematologic diseases. Early diagnosis of infection, rapid identification of the causative pathogen(s), and prompt initiation of appropriate antimicrobial treatment (the first 24 hours are most critical) all have a major impact on mortality.

The LightCycler® SeptiFast Test MGRADE (SeptiFast Test) is an in vitro nucleic acid amplification test for the direct detection and identification of DNA from bacterial and fungal microorganisms in human EDTA whole blood. The SeptiFast test can detect nucleic acids from the most common pathogens (approximately 90%) responsible for hospital-associated bacteremia. The test is used in conjunction with the patient's clinical presentation and established microbiological assays and other laboratory markers as an aid in antimicrobial treatment decision making for patients with suspected sepsis and other bloodstream infections.

This is a randomized prospective study of the use of the SeptiFast Test as an adjunct to traditional management of neutropenic haematological patients suspected of having infection or sepsis. The study will be performed in a two-armed manner. The blood sample for the SeptiFast Test will be collected from all included patients. However, analysis of the SeptiFast Test in the control group will only be performed at a later point in time; thus, in the control group results will not become available until the end of the study and, therefore, cannot be used for guiding clinical decisions.

Patients complete the study when the episode of infection or sepsis resolves, or the patient is discharged from a hospital, or the patient died.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with hematological disease and neutropenia < 500/µl (or < 1000/µl, if criterion 5A is fulfilled)
2. Known or acute infection, or suspected infection, or sepsis, which clinically indicates investigation by blood culture
3. Time-frame after diagnosis or suspicion of infection or sepsis: < 72 hours
4. Species causing infection not known before inclusion
5. Patient fulfils criterion A or/and B

   A. Indication for an initiation of antimicrobial therapy in patients with febrile neutropenia
   * Neutropenia <500/µl or <1000/µl if decline to <500/µl is expected in the next 48h.
   * Single (oral) temperature of ≥ 38.3°C, or temperature ≥ 38.0°C lasting for at least 1h or measured twice within 12h.
   * No evidence of non-infectious cause of fever (blood products, drugs reactions, etc)

   B. At least two of the following criteria:
   * Temperature >38°C or <36°C
   * Heart rate >90 beats/minute
   * Respiratory rate >20 breaths/minute or PaCO2 <32 mmHg / 4,3 kPa
6. Patient is able to provide written informed consent

Exclusion Criteria:

1. Moribund patients with survival expectation < 24h
2. Younger than 18 years
3. Patient is not able to provide informed consent
4. Patients not suitable for study participation in the opinion of investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The number of changes in empirical antimicrobial therapy | up to the end of study participation
Time to the change to the targeted antimicrobial therapy | at time point of change to the targeted antimicrobial therapy

SECONDARY OUTCOMES:
The number of patients with a potential pathogen identified by the SeptiFast Test, compared with the number of patients likely to have bloodstream infection or sepsis, as determined by a constructed clinical comparator | at day 1 and 72h after study inclusion
Number of patients having a change to a more appropriate antimicrobial (evaluated retrospectively by susceptibility) | up to the end of study participation
Time to identification of a potential pathogen | at time point of identification of a potential pathogen
Time to change antimicrobial to a more appropriate antimicrobial | at time point of change to a more appropriate antimicrobial
Duration (in days) of antimicrobials | up to the end of study participation
Change in condition severity (clinical parameters) | daily
Days in intensive care unit (ICU) | at the end of study participation
Ventilation duration in ICU (hours) | at the end of study participation
Days in hospital (from study inclusion) | at the end of study participation
All-cause death | at the end of study participation
Treatment costs | up to the end of study participation

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Becker, MD, Professor, Principal Investigator — Institute of Medical Microbiology, University Hospital Muenster
Locations (1):
- University Hospital Muenster, Münster, North Rhine-Westphalia, Germany